CLINICAL TRIAL: NCT04577313
Title: DOSE DETERMINATION TRIAL: The Start/Persist Studies
Brief Title: HIV Treatment Adherence Dose Determination Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Connecticut (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H19-161; R01MH121129 (NIH)
Record Dates: First submitted 2020-09-23; First posted 2020-10-06 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Continuous Counseling (Active Comparator): Receives up to 16 weekly behavioral counseling sessions over the phone to achieve optimal medication adherence. Counseling adjusts to patient needs and determines the dose to achieve optimal adherence / HIV suppression, in contrast to the fixed dose condition that does not adjust to patient response.
  Interventions: Behavioral: Behavioral Self-Regulation Adherence Counseling
- Fixed Counseling (Active Comparator): Receives up to five weekly behavioral counseling sessions over the phone focused on improving HIV medication adherence / viral suppression.
  Interventions: Behavioral: Behavioral Self-Regulation Adherence Counseling

INTERVENTIONS:
Behavioral: Behavioral Self-Regulation Adherence Counseling — Telephone-delivered counseling to focus on cognitive-behavioral skills to improve HIV treatment adherence.

SUMMARY:
The proposed research will conduct the first dose-determination trial to find the optimal number of behavioral counseling sessions (dose) needed to achieve and sustain optimal HIV treatment adherence. The results of this study will determine how much intervention is needed for whom and at what cost to guide health policy and implementation of behavioral interventions designed to improve durable viral suppression.

DETAILED DESCRIPTION:
The proposed research will conduct the first ever dose-determination trial of a behavioral intervention to improve engagement in HIV care, antiretroviral therapy (ART) adherence and HIV viral suppression. The trial is designed to inform the implementation of behavioral interventions, including several in CDC's Compendium of Evidence-Based Interventions. Behavioral counseling has the flexibility and reach to overcome numerous challenges to HIV care, including social, emotional, and structural barriers. However, basic questions of how to best implement and scale-up interventions remain unanswered, such as "how much intervention is needed to achieve HIV suppression in subgroups of patients facing individual and social challenges?" There are currently no dose-determination trials in the HIV behavioral intervention literature to guide implementation decisions and health service policy. In the proposed research the investigators specifically aim to: (a) determine the minimum effective dose of an evidence-based HIV treatment engagement and adherence intervention, (b) identify subgroups of patients requiring greater and fewer intervention resources to achieve and sustain viral suppression, and (c) the costs associated with intervention dose-response. Participants who are receiving ART with empirically determined low-adherence will be randomized to either: (a) the dose determination condition of weekly evidence-based behavioral self-regulation counseling until achieving HIV suppression or (b) fixed dose 5-weekly sessions of evidence-based behavioral self-regulation counseling sessions. The dose determination condition adjusts to patient needs and determines the dose to achieve optimal adherence / HIV suppression, in contrast to the fixed dose condition that does not adjust to patient response. The trial is therefore designed to determine the number of behavioral counseling intervention sessions needed to achieve and sustain HIV suppression. Once meeting criteria for adherence / viral suppressed, counseling in the dose-determination condition is suspended. In contrast, the fixed-dose condition is delivered in five prescribed sessions as disseminated by the CDC. Follow-up assessments commence for 12-months from baseline with the primary endpoint of 12-month blood plasma HIV viral load and secondary outcome of ART adherence. Response to counseling is defined by achieving viral suppression and non-response is defined by not achieving optimal adherence / viral suppression. Participants in both the dose-determination and fixed-session conditions who initially respond and rebound to unsuppressed viral load will receive additional counseling with redose-response monitored and analyzed. Longitudinal analyses will examine intervention dose for key patient subgroups and dose-response cost-effectiveness analyses to guide resource allocation and implementation decisions. This research is aimed at informing health policy makers and programmatic decisions regarding intervention implementation to increase the likelihood of sustained HIV suppression.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed HIV positive
* Confirmed prescribed antiretroviral therapy
* Confirmed non-adherent to anti-retroviral therapy

Exclusion Criteria:

* Does not have access to a phone
* Does not have access to the internet

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Change in Antiretroviral Therapy Adherence from Baseline to 12-Months | 12-Month
  Medication adherence defined by percentage of medication doses taken as prescribed
Change in HIV Viral Load from Baseline to 12-months | 12-months
  Blood plasma HIV RNA

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Connecticut, Storrs, Connecticut
  - University of Connecticut Field Site, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: No
Data sets masked for all patient level identifying information.

REFERENCES:
- [Background] Kalichman SC, Kalichman MO, Cherry C, Eaton LA, Cruess D, Schinazi RF. Randomized Factorial Trial of Phone-Delivered Support Counseling and Daily Text Message Reminders for HIV Treatment Adherence. J Acquir Immune Defic Syndr. 2016 Sep 1;73(1):47-54. doi: 10.1097/QAI.0000000000001020. PMID 27105048